CLINICAL TRIAL: NCT00650442
Title: Evaluation of the Adhesion Quality and Primary Dermal Irritation Potential of an Alternate Second Generation Estradiol Transdermal Systems in Normal Healthy Female Volunteers
Brief Title: Evaluation of Adhesion Quality and Irritation of an Alternate Second Generation Estradiol Transdermal System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullivan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: ESTR-02133
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Estradiol Transdermal System Placebo - Alternate Adhesive
  Interventions: Drug: Estradiol Transdermal System Placebo - Alternate Adhesive
- 2 (Placebo Comparator): Estradiol Transdermal System Placebo - Current Adhesive
  Interventions: Drug: Estradiol Transdermal System Placebo - Current Adhesive

INTERVENTIONS:
Drug: Estradiol Transdermal System Placebo - Alternate Adhesive — single application
  Arms: 1
Drug: Estradiol Transdermal System Placebo - Current Adhesive — single application
  Arms: 2

SUMMARY:
The primary objective of this study was to compare the adhesive quality of the current Mylan estradiol placebo transdermal system, with that of an alternate second generation Mylan estradiol placebo transdermal system following a single system application. As a secondary objective, primary dermal irritation was assessed after removal of each transdermal system.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-66 years.
2. Sex: Females only.
3. Weight: At least 52 kg (115 lbs) and within 20% of Ideal Body Weight (IBW), as referenced by the Table of ""Desirable Weights of Adults"" from Metropolitan Life Insurance Company, 1999 (See Part II: ADMINISTRATIVE ASPECTS OF HUMAN DERMAL SAFETY STUDY PROTOCOLS).
4. All subjects should be judged normal and healthy during a prestudy medical evaluation (physical examination, laboratory evaluation and 12-lead ECG) performed within 14 days of the initial patch application.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Any prior history of skin diseases (eczema, psoriasis, atopic dermatitis).
3. Damaged skin in or around test sites that include sunburn, uneven skin tones, tattoos, scars or other disfigurations of the test site.
4. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II: ADMINISTRATIVE ASPECTS OF HUMAN DERMAL SAFETY STUDY PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
5. Subjects who have received an investigational drug within 30 days prior to the initial patch application and/or participated in any transdermal system test for irritation or sensitization within the last 4 weeks.
6. Allergy or hypersensitivity to any tapes or adhesives (ex. band-aids, medical tape).

Ages: 40 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Transdermal Adhesion | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Clark, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html